CLINICAL TRIAL: NCT01180101
Title: Effects of Intentional Weight Loss Interventions in Chronic Kidney Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-380
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Kidney Disease; Obesity
Keywords: Obesity; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Obesity | interventions — Diet; Exercise; Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lifestyle modification group (Active Comparator): This group will undergo supervised exercise training 5 days per week and follow hypocaloric diet for 12 weeks. All exercise training sessions will be supervised by an Exercise Physiologist or Research Nurse, and will be conducted in the Exercise Physiology Laboratory at the CCF CRU. Exercise training will consist of walking, running on a treadmill, and stationary cycling on a cycle ergometer. Each exercise session will include a brief standardized warm-up and cool-down that include a series of stretching exercises.
  Interventions: Behavioral: Diet and exercise
- Bariatric Surgery Group (Active Comparator): This group will include CKD patients who undergo bariatric surgery.
  Interventions: Procedure: Bariatric Surgery
- CKD Group (control) (No Intervention): This group will not undergo any form of weight loss intervention

INTERVENTIONS:
Behavioral: Diet and exercise — This group will follow a hypocaloric diet and supervised exercise training for 12 weeks.
  Arms: Lifestyle modification group
Procedure: Bariatric Surgery — Patients will undergo bariatric surgery
  Arms: Bariatric Surgery Group

SUMMARY:
Obesity is an established risk factor for development and progression of kidney disease. Intentional weight loss in people without kidney disease results in an improvement in diabetes, blood pressure, cholesterol, cardiovascular disease and overall death rates. The investigators do not know whether this holds true in patients with chronic kidney disease. In the proposed pilot study, the investigators will analyze if kidney function stabilizes after weight loss interventions in obese kidney disease patients and the mechanisms that might mediate this beneficial effect. If weight loss in kidney disease patients results in stabilization of kidney function, this would provide an opportunity to conduct a long-term prospective study to analyze the sustained benefits of weight loss in kidney disease patients.

Specific aim 1:

To ascertain the effects of lifestyle modification or bariatric surgery on urinary protein excretion and renal function among obese CKD patients.

Hypothesis: Weight loss attained through either lifestyle modification or surgical intervention will result in lowering of urinary protein excretion and stabilization of renal function among obese CKD patients.

Specific aim 2:

To identify the mechanism that mediates the change in urinary protein excretion and renal function among obese CKD patients undergoing lifestyle modification or bariatric surgery.

Hypothesis: Weight loss attained through either lifestyle modification or surgical intervention will result in amelioration of endothelial dysfunction, inflammation, insulin resistance and an increase in High Molecular Weight (HMW) adiponectin levels that then mediate the improvement in urinary protein excretion and renal function among obese CKD patients.

DETAILED DESCRIPTION:
In this non-randomized prospective study, three different groups of patients will be enrolled. Group 1 will include obese chronic kidney disease (CKD) patients undergoing lifestyle modifications, Group 2 will include obese CKD patients undergoing bariatric surgery and Group 3 will include obese CKD patients undergoing no specific weight loss interventions (control group).

The lifestyle group will undergo supervised exercise training 5 days per week and follow hypocaloric diet based on the recommendations by a dietitian for 12 weeks. The exercise training will consist of walking, running on a treadmill and stationary cycling on a cycle ergometer. Patients will undergo adipokines, markers of inflammation,insulin resistance, renal function, bioimpedance analysis,DEXA measurement at baseline, 3- and 6-month intervals. CKD patients who undergo bariatric surgery and the control group will also undergo same blood tests, renal function studies and body composition studies at baseline, 3- and 6-month intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age > 18 years) individuals with BMI > 35 kg/m2
2. Patients with stage III CKD (eGFR 30-59 ml/min and with or without microalbuminuria or proteinuria)
3. Individuals who are eligible for bariatric surgery, based on National Institutes of Health and clinical criteria (BMI > 40 kg/m2 BMI > 35 kg/m2 with co-morbidities and > 18 years of age), and do not have any health related or psychiatric contraindications for the surgery (for bariatric surgery group only)

Exclusion Criteria:

1. History of prior and functioning kidney transplant or on dialysis
2. Cardiovascular conditions including significant known coronary artery disease (recent PCI or CABG within last 6 months), uncompensated congestive heart failure and/or EF <30%, history of stroke (within last 6 months), or uncontrolled hypertension (defined as SBP > 180 mm Hg or DBP > 110 mm Hg).
3. HbA1C >8.0%
4. Hemoglobin <10 g/dl or hematocrit <30 (within the last 6 months)
5. Presence of active inflammatory disease such as AIDS, hepatitis B or C, or other active inflammatory diseases such as vasculitis
6. Patient being treated for malignancy (excluding basal or squamous cell carcinoma of the skin)
7. Patients taking anti-inflammatory medication such as NSAIDS except aspirin < 325 mg/day over the past 30 days, or on any dose of prednisone therapy
8. On other study drug protocols
9. Patient on beta-blocker therapy - only for diet/exercise group
10. Patients can be on Angiotensin converting enzyme inhibitors/Angiotensin receptor blocker therapy that was started at least 3 months prior to the enrollment. New Angiotensin converting enzyme inhibitors/Angiotensin receptor blocker therapy initiation will not be allowed during the study period

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-08; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in renal function using iothalamate studies and urinary protein excretion using 24 hour urinary studies | 6 months
  Weight loss attained through either lifestyle modification or surgical intervention will result in lowering of urinary protein excretion and stabilization of renal function among obese CKD patients.

SECONDARY OUTCOMES:
Changes in markers of insulin resistance and inflammation, adipokines, and body composition. | 6 months
  Weight loss attained through either lifestyle modification or surgical intervention will result in amelioration of endothelial dysfunction, inflammation, insulin resistance and an increase in HMW adiponectin levels that then mediate the improvement in urinary protein excretion and renal function among obese CKD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Sankar Navaneethan, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States